CLINICAL TRIAL: NCT00532987
Title: Assessment of Health Related Quality of Life in Patients Treated for Rectal Cancer
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: REC0003; 79517 (Other: Stanford University Alternate IRB Approval Number); REC0003 (Other: Stanford University)
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Rectal Cancer; Colon Cancer; Anal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Anus Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire form to be completed by patient
  Other Names: Research survey

SUMMARY:
Treatment of rectal cancer often consists of surgical resection of the tumor. Chemotherapy and/or radiotherapy are frequently given before or after surgery. In this study, we wish to learn if there are differences in the treatment effectiveness or in the quality of life of patients based on their type of treatment (e.g. Radiotherapy and chemotherapy before or after surgery). Information from this questionnaire collected from you and other patients may help improve the quality of life of rectal cancer patients in the future. Medical information on your tumor, treatment received, and side effects will be compiled and maintained in a database to learn more about outcomes of treatment for rectal cancer.

DETAILED DESCRIPTION:
There exists little published data studying the health related quality of life (HRQOL) of patients treated for the rectal cancer. Patients are commonly treated with surgery preceded or followed by chemo radiotherapy. Patients chart review and questionnaires administered during follow-up exam or by mailing will be use to compile data comparing the HRQOL of the two study groups(Preoperative versus Post operative chemotherapy).

Our Radiation Oncologist will also informed all the new pts. under going radiotherapy regarding this study and will encourage them in become part of our study population. The prospective study will help us in increasing the number of participants and also it give us an opportunity following the patients as they go through their treatment.

Through the use of department databases, a cohort or rectal cancer patients treated at Stanford will be identified. Patients demographics, treatment received ,disease outcomes, and treatment associated complications will be compiled from available data. HRQOL questionnaires will be answered through a mailing or during clinic visits. Treatment outcomes, toxicities and overall quality of life of preoperative and postoperative chemo radiotherapy treatment group will be compared in relation to the lesion location.

ELIGIBILITY:
Inclusion Criteria:History of histologically-confirmed rectal cancer with treatment or undergoing treatment at Stanford University Hospital.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: History of histologically-confirmed rectal cancer with treatment or undergoing treatment at Stanford University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2003-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lane Welton, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States